CLINICAL TRIAL: NCT03036423
Title: Cognitive Training to Protect Immune Systems of Older Caregivers
Brief Title: Cognitive Training for Older Caregivers
Acronym: CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kathi Heffner, Associate Professor of Nursing and Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY0001991; R01AG049764 (NIH)
Record Dates: First submitted 2016-11-10; First posted 2017-01-30 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Life Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online video education (Active Comparator): Participants will have computer access to a library of videos, including various lectures and demonstrations of interest, from which to select and view.
  Interventions: Behavioral: Online video education
- Computerized mental exercises (Active Comparator): Participants will use a computer to do a variety of activities which are customizable to their own abilities and progress.
  Interventions: Behavioral: Computerized mental exercises

INTERVENTIONS:
Behavioral: Online video education
  Arms: Online video education
Behavioral: Computerized mental exercises
  Arms: Computerized mental exercises

SUMMARY:
The purpose of this study is to test whether certain brain training activities can promote cognitive, emotional, and physical health in caregivers of a loved one with dementia. Numerous studies show that family dementia caregiving can be stressful, and can increase mental and physical health risks. This study aims to understand how to reduce those risks.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking (consent process and assessments will be conducted in English only)
* Currently living with or in proximity to, and the primary caregiver for a loved one with dementia who lives in the community-for the purposes of this study, "loved one" refers to a family member such as a spouse, ex-spouse, significant other, sibling, in-law, parent, or other type of close established relationship (e.g., close friend) regarded as family; "primary caregivers" provide daily informal (non-paid) in-person care.
* Currently experiencing moderate to high levels of perceived stress and caregiver burden. Caregivers will be screened for stress levels and caregiving burden using the 10-item Perceived Stress Scale (PSS 10) and the Modified Caregiver Strain Index (MCSI), respectively. Caregivers scoring above the population mean (approx.) on the PSS 10 (> 11), reporting at least moderate caregiver strain (score ≥ 5) on the MCSI will be eligible for participation.

Exclusion Criteria:

* cognitive impairment or dementia (identified by the Montreal Cognitive Assessment (MoCA)). Cutoff scores on the MoCA will be 23 or lower except for subjects who identify as black or African American, in which case cutoffs will be based on scores from the sample population reported in Rossetti et al (2017); subjects scoring greater than one standard deviation below the published score, by respective age and education, will be excluded.
* current major depression (current Major Depression diagnosis and/or Geriatric Depression Scale (GDS 15) score ≥ 10)
* no recent (within 2 months) major surgery
* History of events that cause neurological injury (e.g., stroke, transient ischemic attack, traumatic brain injury or head injury with loss of consciousness)
* Serious psychiatric or alcohol/substance use disorders, including current alcohol dependence, current non-alcohol psychoactive substance use dependence, psychotic disorders or features (current and lifetime), bipolar disorder (determined from Mini International Neuropsychiatric Exam (MINI) modules)
* Autoimmune disorder (e.g., Crohn's disease, lupus, rheumatoid arthritis)
* Active neoplastic disease or receiving immunosuppressive therapy for cancer (or < 6 months post-chemo or radiation) or other diseases (< 3 months prior to enrollment)
* No significant immunodeficiency disorder (e.g., alymphocytosis, hepatitis B or C, HIV)
* Serious cardiovascular disease (e.g., congestive heart failure, pacemaker) or myocardial infarction within past 6 months
* Physical condition precluding required activities as part of the computerized cognitive training (e.g., inability to use a computer mouse; inadequate visual acuity)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Useful Field of View test performance at 12 months after the intervention | 12 months after the intervention
  Useful Field of View computerized test of speed of processing and attention; lower score (in milliseconds) reflects better performance
Resting high frequency heart rate variability (HF-HRV) at 12 months after the intervention | 12 months after the intervention
  HF-HRV is derived by spectral analysis of the electrocardiograph (ECG) waveform and is a measure of parasympathetic control of the heart; Higher resting HF-HRV (in Hz) reflects greater parasympathetic regulation of the heart
Emotion regulation at 12 months after the intervention | 12 months after the intervention
  Measured as change in negative affect (from responses to the self-assessment manikin on a 9-point scale) from before to after a mental challenge; less increase in negative affect score suggests better emotion regulation
Emotional well-being at 12 months after the intervention | 12 months after the intervention
  The primary index of emotional well-being will be depressive symptoms (Center for Epidemiology Studies Depression scale); a lower score on this measure indicates less depressive symptoms
Immune aging | 12 months after the intervention
  Identified from blood samples; lower levels of inflammation (measured by enzyme-linked immunosorbent assay (ELISA) assay) and T-lymphocyte profiles that reflect larger ratios of naïve T-cells relative to mature T-cells (measured from flow cytometry) will index less aging of the immune system

CONTACTS AND LOCATIONS:
Overall Officials: Kathi L Heffner, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heffner KL, Crean HF, Gallegos AM, Quinones-Cordero MM, Weber MT, Sorensen S, Lin RSY, Podgorski CA, Lin FV. Speed of Processing Training for Stress Adaptation in Caregivers of a Family Member With Dementia: A Randomized Controlled Trial. Innov Aging. 2025 Mar 22;9(5):igaf033. doi: 10.1093/geroni/igaf033. eCollection 2025. PMID 40454426

DOCUMENTS (1):
  • Informed Consent Form (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT03036423/ICF_000.pdf